CLINICAL TRIAL: NCT03264716
Title: A Prospective Open-label Study of Transarterial Chemoembolization by Hepasphere Microspheres for the Treatment of Unresectable Colorectal Liver Metastasis
Brief Title: Transarterial Chemoembolization by Hepasphere Microspheres for the Treatment of Unresectable Colorectal Liver Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201701124DIPB
Record Dates: First submitted 2017-05-11; First posted 2017-08-29 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-06

CONDITIONS: Unresectable Colorectal Liver Metastasis
Keywords: TACE (transarterial chemoembolization); colorectal liver metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HepaSphere TACE (transarterial chemoembolization) (Experimental): Using HepaSphere TACE (transarterial chemoembolization) for colorectal liver metastasis. TACE using HepaSphere load with doxorubicin.
  Interventions: Device: HepaSphere TACE (transarterial chemoembolization)

INTERVENTIONS:
Device: HepaSphere TACE (transarterial chemoembolization) — 100 mg doxorubicin will be loaded onto the HepaSphere Microspheres and delivered via microcatheter.

SUMMARY:
Colorectal cancer is the third most frequently diagnosed cancer and the third leading cause of cancer related deaths in Taiwan. Of the 10,248 new colorectal patients diagnosed each year approximately 60% will develop liver metastasis during the course of their disease. In approximately 30% of these patients who develop liver metastasis the metastatic disease will remain confined to the liver.

For the 70-75% of colorectal patients with colorectal liver metastasis not suitable for hepatic resection or similarly ablative therapy with curative intent, systemic chemotherapy is the standard initial management. However, after a patient has failed first- line and in some cases second-line chemotherapy, response rates fall to as low as 12% (Chen HX 2006). Transarterial chemoembolization (TACE) with microsphere is an alternative treatment because normal liver tissue receives most of its blood supply from the portal vein, while colorectal liver metastases derive most of their flow from the hepatic artery. Several clinical trials have explored the feasibility and the efficacy of TACE with microsphere as a treatment for patients with colorectal liver metastasis. HepaSphere represents a novel drug delivery system for chemoembolization, which can add two benefits to embolization therapy. First, by ionically binding the doxorubicin throughout the microspheres, more drug can be delivered into the tumor, with less escape into peripheral circulation. Second, conformability to the architecture of the vessel lumen, providing more contact surface area with the embolic material and the vessel intima, leading to a more complete occlusion. However, there are limited experiences in using HepaSphere TACE for colorectal liver metastasis in Taiwan. In this pilot study, we will evaluate the initiate safety and efficacy of Hepasphere microspheres loaded with a chemotherapeutic agent doxorubicin for the treatment of patients who have failed first-line and second-line systemic chemotherapy.

DETAILED DESCRIPTION:
This is an open-label, non-comparative study aimed to evaluate the safety profiles and efficacy of patients with unresectable colorectal liver metastases treated by selective TACE (transarterial chemoembolization) using HepaSphere load with doxorubicin. Total of 15 patients will be planned to recruit.

The study procedures will consist of a screening period in which patient eligibility will be determined. Patients meeting the study entry criteria will receive one HepaSphere treatments. Computed tomography (CT) will be done 4 weeks after treatment to determine tumor response.

Hepatic progression free survival will be followed from the date of first study HepaSphere procedure until a date of target liver tumor progression is obtained or the patient is lost to follow-up. Treatments for liver metastases after the study HepaSphere treatments are complete will be documented during the survival period to the extent possible.

The investigators will evaluate subjects' previous treatments and response, and determine to use doxorubicin for subjects. 100 mg doxorubicin will be loaded onto the HepaSphere Microspheres (through ionic bonding when the spheres are exposed to doxorubicin solubilized in non-ionic contrast medium) and delivered via microcatheter. No ethiodized oil is used with the microspheres. The occlusion endpoint will be stasis to the second or third branches. If stasis has not been reached when the target dosage of doxorubicin has been delivered, additional bland embolic agent will be used to achieve a consistent endpoint. Other concurrent chemotherapy, such as Xeloda, 5-fluorouracil but not limited, can be used in combination with HepaSphere Tx.

The study will evaluate safety throughout the protocol specified treatment phase of the investigation by assessing adverse events, as well as changes from baseline in laboratory values, findings on physical examination including vital signs and Eastern Cooperative Oncology Group (ECOG) performance status. Concomitant medication usage will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria in order to be entered into the study:

  1. Liver dominant metastatic colorectal cancer
  2. Metastatic colorectal patients who have failed first-line and second-line systemic chemotherapy.
  3. ECOG 0 to 1 or a Karnofsky Performance score of 80-100%;
  4. Age 20 years or older
  5. Patient has signed informed consent

Exclusion Criteria:

- If patients meet any of the following criteria they may not be entered into the study:

1. History of severe allergy or intolerance to any contrast media not controlled with premedication
2. Severe peripheral vascular disease that would preclude catheterization
3. Significant extra-hepatic disease, generally in excess of 50% of the overall whole body tumor bulk outside the liver, or any tumor burden that represented an imminent threat to the patient's life
4. Greater than 75% hepatic parenchymal involvement. Previous treatment with any form of transarterial embolization for liver tumors

f. Female patients who are pregnant, breastfeeding, or premenopausal and not using an effective method of contraceptive g. Any contraindication to arteriography or hepatic embolization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Hepatic Progression free survival | up to one year
  To define all participants from the day of the first HepaSphere Tx until the date that hepatic progression or death is first reported, whichever comes first.

SECONDARY OUTCOMES:
An overall tumor response classification | up to one year
  The tumor response will be assessed using modified Response Evaluation Criteria In Solid Tumors (mRECIST) criteria to evaluate tumor necrosis, and includes assessment of viable tumor, which is defined as uptake of contrast agent in the arterial phase of computed tomography (CT).

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD. PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No